CLINICAL TRIAL: NCT00509990
Title: Open Label Multicenter Study, 52 Weeks Duration, Using Pimecrolimus Cream 1% for the Long-term Treatment of Mild to Moderate Atopic Dermatitis in Pediatric Patients Within a Usual Clinical Setting
Brief Title: Open Label Study of Long Term Treatment of Pediatric Treatment of Atopic Dermatitis With Pimecrolimus Cream 1% Within a Usual Clinical Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASM981CVE01
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, pimecrolimus, children
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 %
  Other Names: Elidel

SUMMARY:
An open-label, multicenter study, of long term management to evaluate effectiveness, tolerability and safety of pimecrolimus cream 1% in pediatric patients with mild to moderate atopic dermatitis in a daily practice

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 months to 12 years old
* Clinical diagnosis of atopic dermatitis
* History of mild to moderate atopic dermatitis
* Investigator Global Assessment ≥ 1 (almost clear/clear of disease)
* Written informed consent

Exclusion Criteria:

* Investigator Global Assessment ≥ 4 (severe/very severe disease)
* Patients with active skin viral infections (i.e, herpes simplex, herpes zoster, varicella)
* Patients with atopic dermatitis, with active clinical infection on area of disease. All active infections must be treated prior to trial inclusion
* Patients in an Immunosuppressive state or with history of malignant disease
* Patients with clinical conditions other that Atopic Dermatitis that according to the investigator may interfere with the evaluation (i.e, Psoriasis, Netherton Syndrome)
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of pimecrolimus cream 1% in the long-term management in mild to moderate atopic dermatitis in pediatric patients in a daily practice, as assessed by: • Investigator Global Assessment • Facial Investigator Global Ass

SECONDARY OUTCOMES:
• To monitor the safety of pimecrolimus cream 1% in the long-term management as assessed by Adverse Events and Serious Adverse Events collection • To evaluate quality of life of both parent and patient assessed by questionnaire. • To determine ste

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis Pharma AG, Basel, Switzerland
Locations (6):
- Mexico (3):
  - Novartis Investigative Site, México
  - Novartis Investigative Site, Monterrey
  - Novartis Investigative Site, Puebla City
- Venezuela (3):
  - Novartis Investigative Site, Aragua
  - Novartis Investigative Site, Edo, Carabobo
  - Novartis Investigative Site, Caracas